CLINICAL TRIAL: NCT04047342
Title: Assessing the Impact of myHealth Rewards Program-related Communications on New Hire Enrollment
Brief Title: Assessing the Impact of myHealth Rewards New Hire Enrollment Emails
Status: Completed | Type: Observational
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0586
Record Dates: First submitted 2019-07-29; First posted 2019-08-06 (Actual); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Health Promotion; Wellness Programs
Keywords: Prospect theory

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard welcome email: The standard welcome email mentions the benefits of enrollment (maintaining good health and saving money on insurance premiums), the average premium savings, the ease of the registration process, and the deadline for registering and having health measures on file, plus it provides registration steps and hyperlinks for registering and finding free health screenings where health measures can be collected and registered at one convenient time and location.
  Interventions: Behavioral: Welcome email
- Loss frame email: The loss frame email recommends that GHP members not "throw away" a precise dollar amount in savings (over $2,000) by not participating and that they can therefore avoid missing out on substantial gains (i.e., savings) by taking action.
  This intervention frames the status quo as a state from which recipients, via inaction, are slated to forfeit a sizable and precise monetary amount to which they should otherwise feel entitled (via loss aversion and the endowment effect). People tend to be risk-seeking in the domain of losses; therefore, this intervention is hypothesized to increase enrollment in the hope of achieving zero loss by meeting program goals, as opposed to a sure loss via inaction.
  Interventions: Behavioral: Welcome email; Behavioral: Loss frame

INTERVENTIONS:
Behavioral: Welcome email — Email
Behavioral: Loss frame — Email
  Other Names: Endowment effect
  Groups: Loss frame email

SUMMARY:
The purpose of the study is to evaluate, prospectively, the potential impact, on myHealth Rewards wellness program enrollment prior to the 2019 November submission deadline, of sending different messages via email to Geisinger Health Plan (GHP) members who have just been hired.

DETAILED DESCRIPTION:
The myHealth Rewards wellness program managed by GHP rewards those GHP members who carry their insurance through employment at Geisinger with reduced health insurance premiums over the course of the following year, if members register for the program and have their health measures on file by the enrollment deadline and are then able to meet their health goals by the respective due date. In spite of the potential savings to health plan members and the wellness program's potential to motivate engagement in healthy activities (with consequent improvement in health outcomes), about 23% of eligible existing GHP members did not enroll during the primary 2019 enrollment period, even after receiving promotional email communications and reminders. Therefore, the current study was developed to test whether a revised version of a standard welcome email is more effective than the standard email in increasing myHealth Rewards login and enrollment rates. The standard welcome email is what would typically be sent by GHP to encourage enrollment among new hires; it mentions the benefits of enrollment (maintaining good health and saving money on insurance premiums), the average premium savings, the ease of the registration process, and the deadline for registering and having health measures on file, plus it provides registration steps and hyperlinks for registering and finding free health screenings where health measures can be collected and registered at one convenient time and location. The loss frame email recommends that GHP members not "throw away" a precise monetary amount in savings by not participating and that they can therefore avoid missing out on substantial gains (i.e., savings) by taking action. It is hypothesized that, on average, the loss frame email will increase enrollment compared with the standard email, among this population of new hires for whom this is only the second time that they have been informed about myHealth Rewards. Findings will help inform how best to increase enrollment in a wellness program among health plan members who are new to the system.

ELIGIBILITY:
Inclusion Criteria:

* Any Geisinger new hire, regardless of benefits status, who started on or after July 1, 2019 and before November 30, 2019

Exclusion Criteria:

* Existing Geisinger employees hired prior to July 1, 2019
* New hires who do not have an email address on file

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population consists of new Geisinger Health Plan members who are benefits subscribers.
Sampling Method: Probability Sample
Enrollment: 824 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings. The PI did not examine or analyze any data from this study prior to this registration.
Supporting Information: Study Protocol
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

RESULTS

PARTICIPANT FLOW:
Recruitment Details: New employees received emails from July 16, 2019 to October 8, 2019. Enrollment data was gathered until December 20, 2019.
Pre-assignment Details: 7 employees were excluded from analysis, as they registered before the emails were sent (e.g., after learning about the program during new hire orientation).
Groups:
- Standard Welcome Email: The standard welcome email mentions the benefits of enrollment and the deadline for registering and having health measures on file, plus it provides registration steps and hyperlinks for registering and finding free health screenings.
  Welcome email: Email
- Loss Frame Email: The loss frame email recommends that Geisinger Health Plan (GHP) members not "throw away" a precise dollar amount in savings (over $2,000) by not participating and that they can therefore avoid missing out on substantial gains (i.e., savings) by taking action.
  Welcome email: Email
  Loss frame: Email
Period: Overall Study
Arm/Group | Standard Welcome Email | Loss Frame Email
Started | 409 | 415
Completed (We did not receive information on bounced emails, so we assumed that all participants in the data set started and completed the study.) | 409 | 415
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline outcome measure was not applicable, since enrollment and login in response to the email was the outcome. There was no previous email, and participants were selected for not having enrolled in the year of the study period.
Groups:
- Loss Frame Email: The loss frame email recommends that GHP members not "throw away" a precise dollar amount in savings (over $2,000) by not participating and that they can therefore avoid missing out on substantial gains (i.e., savings) by taking action.
  Welcome email: Email
  Loss frame: Email
- Total: Total of all reporting groups
Arm/Group | Standard Welcome Email | Loss Frame Email | Total
Number analyzed (Participants) | 409 | 415 | 824
Age, Categorical [Count of Participants; unit: Participants] — Population: Data were not collected.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data were not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 409 | 415 | 824

OUTCOME MEASURES:

1. Primary Outcome: Number of People Enrolled Within 7 Days
Description: Enrollment in the myHealth Rewards program (yes/no) within 7 full days of the beginning of the intervention for each cohort (i.e., when the emails are first sent within each weekly new hire cohort). Data will be aggregated across cohorts, including the July 16 cohort and every subsequent cohort through the week prior to reminder emails scheduled to be sent out in October, 2019.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Welcome Email | Loss Frame Email
Number analyzed (Participants) | 409 | 415
Participants | 131 | 130
Statistical Analysis 1: Comparison: Standard Welcome Email vs Loss Frame Email; Test type: Superiority; p = .828, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.72 to 1.30]

2. Primary Outcome: Number of People Who Logged in to the Program Within 7 Days
Description: Logging into the myHealth Rewards program (yes/no) within 7 full days of the beginning of the intervention for each cohort (i.e., when the emails are first sent within each weekly new hire cohort). Data will be aggregated across cohorts, including the July 16 cohort and every subsequent cohort through the week prior to reminder emails scheduled to be sent out in October, 2019.
Time Frame: 7 days
Population: This data was not collected due to administrative error.
Arm/Group | Standard Welcome Email | Loss Frame Email
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No adverse events were evaluated.
Description: We only received aggregate information about email engagement with no individual-level information collected (including those for adverse events).
Arm/Group | Standard Welcome Email | Loss Frame Email
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
For this study, we only received data about engagement with the email (specifically, only enrollment). Individual patients were not identified and demographic information such as age, sex, or gender were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT04047342/Prot_SAP_000.pdf